CLINICAL TRIAL: NCT04186325
Title: Ultrasound Assessment of Diaphragmatic Muscle Exercise in Mechanically Ventilated Patients.
Brief Title: Diaphragm Training Ultrasound
Acronym: DiaphUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: diaphragm ultrasound
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: DIAPHRAGM -Ultrasound -Weaning -Mechanical Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (No Intervention): Group C: the regular mechanical ventilation protocol will be followed.
- Group T (Experimental): Group T: inspiratory muscle training (IMT) will be initiated starting from the first ICU day. IMT will be conducted for 10 minutes two sessions per day, with an initial load of 30% of the maximum inspiratory pressure (MIP) measured immediately after changing patients to pressure support mode, and increased up to 40% in the second 5 minutes if tolerated by the patient. In addition, these patients received the usual care of MV patients.
  Interventions: Procedure: DIAPHRAGMATIC exercising

INTERVENTIONS:
Procedure: DIAPHRAGMATIC exercising — inspiratory muscle training (IMT) will be initiated starting from the first ICU day. IMT will be conducted for 10 minutes two sessions per day, with an initial load of 30% of the maximum inspiratory pressure (MIP) measured immediately after changing patients to pressure support mode, and increased up to 40% in the second 5 minutes if tolerated by the patient. In addition, these patients received the usual care of MV patients.
  Arms: Group T

SUMMARY:
Common neurological indications of intubation and initiation of mechanical ventilation (MV) include ischemic and hemorrhagic stroke, neurotrauma, and intracranial hemorrhage. Mechanical ventilation is frequently applied to protect the airway from the risk of aspiration and to prevent both hypoxemia and hypercapnia, which are two major systemic factors of secondary brain insult.

Mechanical ventilation after endotracheal intubation predisposes these patients to an increased incidence of pulmonary complications such as ventilator-associated pneumonia (VAP), increased risk of deep vein thrombosis, bedsores, increased hospital stay, and poor clinical outcome.

The weaning process from MV involves the reduction of ventilator parameters and Extubation. Daily, careful evaluation of clinical and neurological conditions and completion of spontaneous breathing trial (SBT) should be considered in order to recognize and facilitate the process of withdrawal of the MV.

The diaphragm which is the principal respiratory muscle provides nearly 75% of the resting pulmonary ventilation. However, In ICU patients, the diaphragm is vulnerable to damage from hypotension, hypoxia, and sepsis. Diaphragmatic dysfunction and atrophy is the main precipitating factor for difficult and successful weaning.

ELIGIBILITY:
Inclusion Criteria:

* patients attached to mechanical ventilation will be included in the study after the informed consent of the legal guardian.

Exclusion Criteria:

* Patients with severe acute lung injury, morbid obesity, chest wall deformity, direct diaphragmatic injury, cervical spine and patients who require neuromuscular infusion will be excluded from the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-12-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of diaphragmatic muscle atrophy | seven mechanical ventilation days

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University-Emergency hospital-ICU, Al Mansurah, Egypt